CLINICAL TRIAL: NCT05916404
Title: Investigation of the Effects of Upper Extremity Aerobic Exercise Training on Oxygen Consumption, Muscle Oxygenation and Physical Activity in Patients With Interstitial Lung Disease
Brief Title: Effects of Upper Extremity Aerobic Exercise Training in Patients With Interstitial Lung Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Study director, PT, PhD, Prof.Dr. Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Head of Cardiopulmonary Rehabilitation Clinic, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Gazi University-58
Record Dates: First submitted 2023-04-29; First posted 2023-06-23 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Interstitial Lung Disease
Keywords: Interstitial Lung Disease; Upper Extremity; Aerobic Exercise; Oxygen Consumption; Physical Activity
MeSH Terms: conditions — Lung Diseases, Interstitial; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple-blind study; the patients will not be informed about their groups (training group or the control group) and they will be evaluated and trained at different places and times.
  Evaluations and interventions will be performed different physiotherapist. In addition, before statistical analysis patients' groups will be coded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): The training group will receive upper extremity high-intensity interval aerobic exercise training on an arm ergometer accompanied by a physiotherapist for 6 weeks.
  Interventions: Other: Upper extremity high-intensity interval aerobic exercise training
- Control Group (Sham Comparator): The control group will not be given any training for 6 weeks during the study period.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Upper extremity high-intensity interval aerobic exercise training — High-intensity interval aerobic exercise training will be given to the training group on an arm ergometer 3 days in a week and 30-45 minutes a day for 6 weeks with the assistance of a physiotherapist. The training workload of the active phase of high-intensity interval aerobic exercise training will be applied at 80-100% of peak oxygen consumption or 85-95% of peak heart rate. The training workload of the active recovery phase of high-intensity interval aerobic exercise training will be applied at 50-60% of peak oxygen consumption or 60-75% of peak heart rate.
  In case of desaturation (<90%) during the training in the patients in the training group, O2 support with a nasal cannula will be given to the patient.
  Arms: Training Group
Other: Control Group — The control group will not be given any training during the 6-week period. After the study, the treatment applied to the training group will also be applied to the control group in order to ensure that the patients in the control group are not ethically deprived of rehabilitation.
  Arms: Control Group

SUMMARY:
Severe dyspnea, cough, fatigue, restrictive type ventilation disorder, decreased pulmonary function, impaired gas exchange, decreased cardiovascular function and exercise intolerance are frequently encountered findings in patients with interstitial lung disease. It was demonstrated exercise training has beneficial effects in patients with interstitial lung disease. However, no study investigated the effects of upper extremity aerobic exercise training on outcomes in patients with interstitial lung disease.

DETAILED DESCRIPTION:
Interstitial lung diseases (ILD) are a heterogeneous group of diseases that cause significant mortality and morbidity worldwide. As a result of the chronic inflammatory process in this disease, structural and mechanical pulmonary disorders develop, which are considered the main causes of deterioration in cardiopulmonary functions. Interstitial lung patients have a decrease in both static and dynamic lung volumes and carbon monoxide diffusing capacity (DLCO). As a result of this pathological mechanism, effort dyspnea and an increase in exercise intolerance occur. Therefore, individuals with ILD tend to avoid activities that increase shortness of breath, resulting in decreased physical activity levels and an increased sedentary lifestyle. Individuals whose functional exercise capacities are also limited due to this vicious circle become more dependent in their daily living activities. In addition, peripheral muscle dysfunction is another important factor that causes exercise intolerance in individuals with all chronic lung diseases, including ILD. One of the most important mechanisms triggering peripheral muscle dysfunction in ILD is hypoxia which develops with desaturation. Hypoxia, which causes an increase in oxidative stress, is one of the factors that can cause muscle dysfunction. It has been reported that upper extremity exercise capacity and functional performance are low in individuals with advanced ILD, and it has been stated that upper extremity exercise training may be beneficial in these patients.

However, the effects of upper extremity aerobic exercise training have not been investigated in the literature in patients with ILD. In this context, the primary aim of our study is to investigate the effects of upper extremity interval aerobic exercise training applied to patients with ILD on oxygen consumption, muscle oxygenation, and physical activity level. The secondary aim of the study is to determine the effects of this training on upper extremity functional exercise capacity, respiratory functions, pulmonary diffusion capacity, respiratory and peripheral muscle strength, inspiratory muscle endurance, dyspnea, fatigue, quality of life, sleep quality, anxiety, and depression. For this purpose, our study was planned as a randomized, controlled, three-blind (investigators, patient, and analyzer) prospective study. According to the block randomization result, at least 21 patients with a diagnosis of ILD will be included in the training and control groups.

The training group will be given upper extremity interval aerobic exercise training with arm ergometer for 30-45 minutes 3 days a week for 6 weeks, and the control group will not be given any training during the study. After the study, the treatment applied to the training group will also be applied to the control group in order to ensure that the patients in the control group are not ethically deprived of rehabilitation.

All assessments will be completed in two days, before and after six weeks of training.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ILD according to ATS/ERS criteria,
* Aged between 18-75 years,
* No pulmonary infection during the last month,
* Patients who volunteer to participate in the study

Exclusion Criteria:

Patients with,

* Body mass index >35 kg/m2,
* An acute pulmonary exacerbation within the last 4 weeks, have an acute upper or lower respiratory tract infection,
* Presence of obstructive pulmonary disease,
* Serious neurological, neuromuscular, orthopedic, or other diseases affecting physical functions,
* Participated in a planned exercise program within the last three months,
* Cognitive impairment that causes them to have difficulty understanding and following exercise test instructions,
* Contraindications for exercise testing and/or exercise training according to the American College of Sports Medicine
* Cancer, renal or hepatic diseases,
* Aortic stenosis, complex arrhythmia, with aortic aneurysm,
* Uncontrolled hypertension, diabetes mellitus, heart failure, arrhythmia and serious cardiovascular disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Oxygen consumption | through study completion, an average of 2 year
  Maximal exercise capacity will be assessed with symptom limited cardiopulmonary exercise test on a treadmill at a progressively increasing speed and grade. Oxygen consumption will be measured during the test.
Muscle oxygenation | through study completion, an average of 2 year
  Before the cardiopulmonary exercise test and the 6-minute pegboard and ring test (6-PBRT), during and after the tests the muscle oxygenation will be measured by using a near-infrared spectroscopy device. Oxygenation of the quadriceps muscle during the cardiopulmonary exercise test, and deltoid muscle during the 6-PBRT will be evaluated. For this purpose, the sensor will be placed at the midpoint of the dominant side muscles.
Physical activity level | through study completion, an average of 2 year
  Physical activity level will be evaluated with a multi-sensor activity device. Multisensor metabolic holter device by detecting the three-dimensional movements of patients; It provides data on total energy expenditure (joules/day), active energy expenditure (joules/day), physical activity duration (min/day), average MET (MET/day), number of steps (steps/day), time spent lying down (min/day). The device will be attached to the non-dominant arms of the patients, and they will be told to wear it for 5 consecutive days, remove the device only during the bath, and reinsert it in the same area after the bath. The average of the parameters of the current four days will be taken and analyzed with the "BodyMedia SenseWear® 7.0 Software" program using the age, gender, body weight and height information of the patients.

SECONDARY OUTCOMES:
Respiratory muscle strength | through study completion, an average of 2 year
  Respiratory muscle strength will be assessed with mouth pressure device. Maximal inspiratory and expiratory pressure (MIP and MEP) will be measured during the test. This values is expressed in centimeters of water (cmH2O) and as a percentage (%) of the expected value.
Peripheral muscle strength | through study completion, an average of 2 year
  Shoulder flexion and abduction muscles and Quadriceps femoris muscle strength will be measured by using a hand-held dynamometer. This values is expressed in Newtons (N) and as a percentage (%) of the expected value.
Upper extremity functional exercise capacity | through study completion, an average of 2 year
  6-minute pegboard and ring test will be performed to assess upper extremity functional exercise capacity. As a result of the test, the total number of ring inserted end of six minutes will be recorded in pieces. It will be expressed as a percentage (%) of the expected value. The presence of any symptoms during the test, supplemental oxygen support, and assistive device usage status will be recorded.
Dyspnea perception | through study completion, an average of 2 year
  "Modified Medical Research Council" dyspnea scale will be used to question dyspnea perception during activities. This scale is a 5-point scale based on rating various physical activities that increase shortness of breath. The lowest and highest values on this scale are as follows: Level 0 "No shortness of breath except strenuous exercise" and level 4 "Too breathless to leave the house or breathless while dressing or undressing."
  The London Chest Activity of Daily Living scale (Turkish version) will be used to evaluate dyspnea perception during activities of daily living in patients. The scale has a total of 4 subheadings and a total of 15 items, including personal care (4 items), household chores (6 items), physical (2 items) and leisure (3 items). Each item is scored on a scale of 0-5 points. Sub-title score and total score are evaluated. The total score is a maximum of 75. As the overall score increases, so does the dependence on activities of daily living.
Fatigue | through study completion, an average of 2 year
  Fatigue will be assessed with Fatigue Severity Scale (Turkish version). This scale includes 9 items and each item scores from 1 (strong disagreement) to 7 (strong agreement) point. Fatigue Severity Scale total score is calculates by deriving an arithmetic mean. Cut-score of over 4 means significant fatigue and higher score indicates more severe fatigue.
Life Quality | through study completion, an average of 2 year
  Quality of life will be assessed with Saint George Respiratory Questionnaire (SGRQ) (Turkish version). This questionnaire is a questionnaire used to evaluate the quality of life in respiratory diseases. The questionnaire consists of 3 parts: symptoms (8 items), activities (16 items), effects of the disease (26 items) and a total of 50 items: 3 parts of the test are scored separately. Then the total score is obtained. The total score ranges from 0-100. A score of zero is normal, while a score of 100 represents maximum disability. As the total score increases, it indicates that poor quality of life. In this questionnaire, a change of 4 points with treatment is considered significant.
Sleep Quality | through study completion, an average of 2 year
  The Pittsburgh Sleep Quality Index (Turkish version) will be used to evaluate the sleep quality of the patients. 19 of the questions in the index, which consists of a total of 24 questions, are questions that the individual answers by evaluating himself/herself. The remaining 5 questions are answered by the individual's bed partner or roommate, if any. The questionnaire includes questions asked under 7 main headings: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping medication, and daytime functions. Each of these 7 main headings is first evaluated in its own right. The scores of the 7 components are then summed up. If the total score is above 5 points, it is considered bad sleep.
Anxiety and Depression | through study completion, an average of 2 year
  Hospital Anxiety and Depression Scale (Turkish version) will be used to evaluate the anxiety and depression levels of the patients. It consists of two subdivisions: Anxiety (HAD-A) and depression (HAD-D). 7 questions consisting of odd numbers (questions 1, 3, 5, 7, 9, 11, 13) measure anxiety, and 7 questions consisting of even numbers (questions 2, 4, 6, 8, 10, 12, 14) measure depression. For the answers to each question, a score of 0-3 is made in the form of a quadruple likert. The lowest score that can be obtained from both subscales is 0 and the highest score is 21. As the score increases, the severity of anxiety and depression increases. 0-7 is considered normal, 8-10 is borderline, 11 and above is considered abnormal. 10 points and above for anxiety and 8 points and above for depression are considered significant.
Modified Borg scale | through study completion, an average of 2 year
  The assessment of dyspnea and fatigue perception in all patients at rest, during, and after exercise training will be performed with the Modified Borg scale. In addition, the perception of dyspnea and fatigue before, during, and after the cardiopulmonary exercise test and 6 minutes of pegboard and ring test will be evaluated with the Modified Borg scale. The modified Borg scale is a subjective scale and scores patients' dyspnea at rest and/or during activity on a scale of 0-10. The lowest score of 0 (zero) indicates "not at all" and the highest score of 10 (ten) indicates "very very serious" shortness of breath or fatigue.
Energy expenditure | through study completion, an average of 2 year
  Energy expenditure during the cardiopulmonary exercise test and 6-minute pegboard and ring test will be evaluated with a multi-sensor activity device. It is expressed in joules.
Inspiratory muscle endurance | through study completion, an average of 2 year
  Inspiratory muscle endurance will be measured incremental threshold loading test, in which patients started an initial load of 30% of maximal inspiratory pressure and test load will be increased with among 10% of maximal inspiratory pressure every 2 minutes.
Forced expiratory volume exhaled in the first second (FEV1) | through study completion, an average of 2 year
  Forced expiratory volume exhaled in the first second (FEV1) will be evaluated by using spirometry. FEV1 is the expiratory volume in the first second of an FVC maneuver which is the volume delivered during an expiration made as forcefully and completely as possible starting from full inspiration. FEV1 is expressed in liters (L) and as a percentage (%) of the expected value.
Forced vital capacity (FVC) | through study completion, an average of 2 year
  Forced vital capacity (FVC) will be evaluated by using spirometry. FVC is the volume delivered during an expiration made as forcefully and completely as possible starting from full inspiration. It is expressed in liters (L) and as a percentage (%) of the expected value.
FEV1/FVC ratio | through study completion, an average of 2 year
  This value is the ratio of forced expiratory volume in one second (FEV1) to forced vital capacity (FVC). FEV1/FVC ratio will be evaluated by using spirometry. It is expressed as a percentage (%) of the expected value.
Peak expiratory flow (PEF) | through study completion, an average of 2 year
  Peak expiratory flow (PEF) is the highest flow achieved from a maximum forced expiratory maneuver started without hesitation from a position of maximal lung inflation. PEF will be evaluated by using spirometry. It is expressed in liters (L) and as a percentage (%) of the expected value.
Forced mid-expiratory flow rate (FEF25-75%) | through study completion, an average of 2 year
  Forced mid-expiratory flow rate (FEF25-75%) will be evaluated by using spirometry. FEF25-75% value is forced expiratory flow over the middle one-half of the FVC. It refers the average flow from the point at which 25% of the FVC has been exhaled to the point at which 75% of the FVC has been exhaled. It is expressed in liters (L) and as a percentage (%) of the expected value.
Diffusion capacity for carbon monoxide (DLCO) | through study completion, an average of 2 year
  Carbon monoxide diffusing capacity of the lung (DLCO) is a measurement to assess the lungs' ability to transfer gas from inspired air to the bloodstream. Its measurement uses carbon monoxide to calculate the pulmonary diffusion capacity. The most common method is the standard single-breathe diffusing capacity test. It is expressed in mmol/(min*kPa) and as a percentage (%) of the expected value.
Carbon monoxide transfer coefficient (KCO=DLCO/Va) | through study completion, an average of 2 year
  KCO is CO transfer coefficient, usually written as DLCO/Va, which indicates the efficiency of CO transfer by alveoli. In other words, it is the diffusion capacity of carbon monoxide for each unit of the alveolar volume. The most common method is the standard single-breathe diffusing capacity test. It is expressed in mmol/(min*kPa*L) and as a percentage (%) of the expected value.
Alveolar ventilation (Va) | through study completion, an average of 2 year
  Alveolar ventilation is amount of contributing alveolar units measured by tracer gas. It expressed in liters (L).

CONTACTS AND LOCATIONS:
Overall Officials: Nazire Nur YILDIZ, M.Sc., Study Chair — Gazi University; Meral BOŞNAK GÜÇLÜ, Prof. Dr., Study Director — Gazi University; Riad BEJTA, Pt., Principal Investigator — Gazi University; Nilgün YILMAZ DEMİRCİ, Assoc. Prof., Principal Investigator — Gazi University
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No